CLINICAL TRIAL: NCT00397072
Title: Phase II Study: Systemic Treatment With iv ZK219477-Epothilone in Recurrent Glioblastoma Patients
Brief Title: Epothilone in Recurrent Glioblastoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Principal Investigator, Antonio Silvani, MD, Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZK219477IV
Record Dates: First submitted 2006-11-07; First posted 2006-11-08 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Glioblastoma
Keywords: Glioblastoma recurrent,temozolomide, epothilone
MeSH Terms: conditions — Glioblastoma

ARMS (1):
- ZK-EPO (Experimental): administered iv for 3 h every 21 days; dose reductions to 12 or 9 mg/m2 ZK-EPO were allowed in order to manage any treatment-related toxicity.
  Interventions: Drug: ZK 219477

INTERVENTIONS:
Drug: ZK 219477

SUMMARY:
The purpose of this single arm phase II study is to evaluate safety and efficacy of ZK 219477 in the treatment of temozolomide pre-treated, recurrent GBM patients.

DETAILED DESCRIPTION:
Malignant gliomas remain among the most devastating cancers, and especially for recurrent GBM no standard treatment has been established to date.

ZK 219477 is a fully synthetic analogue of Epothilone B, a naturally occurring cytotoxic substance. ZK 219477 inhibits microtubule depolymerization, causing cell cycle blockage in G2/M phase and induction to apoptosis. This mechanism of action is similar to that of taxanes (paclitaxel and docetaxel), but epothilones retain activity against multi-drug resistance (MDR) tumours. ZK 219477 demonstrated both in vitro and in vivo considerable anti-tumour activity against a wide range of malignancies, and it is now about to enter phase II studies in a number of selected indications. In pre-clinical model ZK 219477 has demonstrated anti-tumorigenic activity for gliomas tumours both in vitro and in vivo.

ZK 219477 has the ability to cross the blood-brain barrier, a fundamental characteristic for a potential GBM chemotherapy. In a preclinical PK study, similar concentrations of ZK 219477 were detected in plasma (1.2 μg/ml) and brain (0.9 μg/g) after 10 min after i.v. application in scid mice. The AUC brain/AUC plasma was about 0.8, indicating a free access to the brain (Hoffmann J et al. 2004, European Journal Cancer Supplement 2, N 8, p. 159, Abstract 521, ref.17). ZK 219477 produced strong antiproliferative activity in the human glioma cell line U373 inoculated subcutaneous in nude mice (2 mg/kg and 9 mg/kg) as well as paclitaxel (8 mg/kg), but on the contrary of paclitaxel, only ZK 219477 demonstrated antitumour activity against U373 implanted in nude mice (9 mg/kg): 8 complete response out 9 treated mice.

Of interest for GBM indication, ZK 219477 is not metabolized by liver cytochrome P450, which is induced by phenytoin and other anti-convulsion drug, commonly used in post-surgery GBM patients.

The purpose of this single arm phase II study is to evaluate safety and efficacy of ZK 219477 in the treatment of pre-treated, recurrent GBM patients. Aim of the study: The purpose of this single arm phase II study is to evaluate safety and efficacy of ZK 219477 in the treatment of pre-treated, recurrent GBM patients. An optional PK study will be performed in selected patients.

Study Design: Open, monocentric, not randomised, single arm, phase II study. Study medication: ZK 219477 epothilone B analog. Study Population: 15 recurrent glioblastoma patients previously treated by surgery, conventional radiotherapy and chemotherapy with temozolomide (TMZ. The 15 patients for this study, represent the first stage of recruitment according to the statistical design.

Inclusion Criteria:

* Histologically proven (at diagnosis) GBM
* Age between 18 and 70 years
* KPS ≥ 70
* Life expectancy of at least 3 months
* Presence of at least one bi-dimensionally measurable lesion on gadolinium (Gd)-enhanced MRI, indicating progressive or recurrent disease at least 8 weeks after standard external-beam radiotherapy
* Recurrence or progression after treatment with radiotherapy and temozolomide. Also patients with residual disease after surgery for recurrent GBM will be included
* Adequate bone marrow reserve (leukocytes ≥ 3,500/ml, ANC ≥ 1,500/ml, platelets ≥100,000/ ml); normal baseline liver (serum bilirubin ≤ 20 /mol/ L), renal (serum creatinine <150 /mol/L) and cardiac function
* Absence of infectious disease, debilitating chronic diseases, and known psychiatric disorders
* Corticosteroid dose stable for at least 1 week
* Adequate recovery from previous surgery, radiation and chemotherapy
* Negative pregnancy test at enrolment in females of child-bearing potential
* Agreement to use highly effective contraception methods in adults of reproductive potential
* Fully informed written consent

Exclusion Criteria:

* Pregnant women
* Patients who have had chemotherapy or radiotherapy within 4 weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZK219477
* Uncontrolled inter current illness including, but not limited, to ongoing or active infection, symptomatic congestive heart failure,unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-infection
* Any prior treatment with epothilones, other tubulin-targetting as taxanes (e.g. paclitaxel, docetaxel) and vinca alkaloids (e.g.vincristine, vinblastine, vinorelbine)
* Peripheral neuropathy
* Any concurrent malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix
* Active infection
* Breast-feeding
* Subjects who have received an experimental drug or have participated in a clinical trial within 3 months prior to screening
* Employees of the investigator or study centre with direct involvement in the proposed study or other studies under the direction of that investigator or study centre

Treatments:

Treatment will be administered on an inpatient basis. ZK 219477 will be administered as an i.v. infusion of 3 hours duration at a dose of 16 mg/m2 BSA every three weeks.

Two dose reductions are allowed in order to manage toxicities: 12 mg/m2 and 9 mg/m2.

Evaluation criteria:

Efficacy evaluation. Primary end-point: Progression Free Survival at 6 months (PFS-6). Secondary end-points: Response rates (CR +PR), Median Survival Time (MST). Safety evaluation. Treatment toxicity will be assessed using CTCAE, Version 3.0, except for neurological toxicity that will be assessed also by means of the Scottish Gynaecological Cancer Trials Group (SGCTG) Neurotoxicity Score and electromyography.

Statistics:

A group-sequential design will be used with the chance of remaining alive and free of progression at 6 months, called "response", as primary endpoint. The null hypothesis of a response rate ≤ 10% will be tested based on the binomial distribution of the response endpoint at a nominal significance level of 0.10 (one-sided). If the observed response rate in the 15 patients is < 20%, the null hypothesis will be accepted and study failure will be concluded. If the observed response rate is ≥ 20% (i.e., at least three out of the 15 patients show a response after 6 months), then consideration would be given to studying further. If the observed response rate amounts to at least 5 out of the initial 15 patients, the null hypothesis will be rejected and the study may be stopped after the first stage. Secondary end-points: PFS and MST will be estimated using the Kaplan-Meier method.

Response, age, KPS, number of surgical procedures performed, previous low grade, and time between end of radiotherapy and start of chemotherapy will be considered variables possibly related to TTP and the time interval between start of chemotherapy and death from any cause (MST). Descriptive statistics with these classified time-to-event variables as subgroups will be provided

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* KPS ≥ 70
* Life expectancy of at least 3 months
* Presence of at least one bi-dimensionally measurable lesion on gadolinium (Gd)-enhanced MRI, indicating progressive or recurrent disease at least 8 weeks after standard external-beam radiotherapy
* Recurrence or progression after treatment with radiotherapy and temozolomide. Also patients with residual disease after surgery for recurrent GBM will be included
* Adequate bone marrow reserve (leukocytes ≥ 3,500/ml, ANC ≥ 1,500/ml, platelets ≥100,000/ ml); normal baseline liver (serum bilirubin ≤ 20 /mol/ L), renal (serum creatinine <150 /mol/L) and cardiac function
* Absence of infectious disease, debilitating chronic diseases, and known psychiatric disorders
* Corticosteroid dose stable for at least 1 week
* Adequate recovery from previous surgery, radiation and chemotherapy
* Negative pregnancy test at enrolment in females of child-bearing potential
* Agreement to use highly effective contraception methods in adults of reproductive potential
* Fully informed written consent

Exclusion Criteria:

* Pregnant women
* Patients who have had chemotherapy or radiotherapy within 4 weeks
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZK219477
* Uncontrolled inter current illness including, but not limited, to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* HIV-infection
* Any prior treatment with epothilones, other tubulin-targetting as taxanes (e.g. paclitaxel, docetaxel) and vinca alkaloids (e.g. vincristine, vinblastine, vinorelbine)
* Peripheral neuropathy
* Any concurrent malignancy other than non-melanoma skin cancer or carcinoma in situ of the cervix
* Active infection
* Breast-feeding
* Subjects who have received an experimental drug or have participated in a clinical trial within 3 months prior to screening
* Employees of the investigator or study centre with direct involvement in the proposed study or other studies under the direction of that investigator or study centre

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival at six months (PFS-6). | 6 months

SECONDARY OUTCOMES:
Response rates (CR +PR) | 2 years
  Secondary end-points
Safety evaluation according to CTC-AE | 2 years
Median Survival Time (MST) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Amerigo Boairdi, MD, Principal Investigator — Istituto Nazionale Neurologico Carlo Besta
Locations (1):
- Istituto Nazionale Neurologico, Milan, Italy

REFERENCES:
- [Background] Klar U, Buchmann B, Schwede W, Skuballa W, Hoffmann J, Lichtner RB. Total synthesis and antitumor activity of ZK-EPO: the first fully synthetic epothilone in clinical development. Angew Chem Int Ed Engl. 2006 Dec 4;45(47):7942-8. doi: 10.1002/anie.200602785. No abstract available. PMID 17006870
- [Result] Silvani A, Gaviani P, Fiumani A, Scaioli V, Lamperti E, Eoli M, Botturi A, Salmaggi A. Systemic sagopilone (ZK-EPO) treatment of patients with recurrent malignant gliomas. J Neurooncol. 2009 Oct;95(1):61-64. doi: 10.1007/s11060-009-9890-8. Epub 2009 Apr 21. PMID 19381446